CLINICAL TRIAL: NCT02216383
Title: Intramuscular Oxytocics: A Randomised Control Trial of Intramuscular Carbetocin, Syntocinon and Syntometrine for the Third Stage of Labour Following Vaginal Birth
Brief Title: Intramuscular Oxytocics: A Randomised Control Trial
Acronym: IMox
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: North Bristol NHS Trust (Other)
Collaborators: Ferring Pharmaceuticals (Industry); University of Bristol (Other); University of the West of England (Other); Royal United Hospital Bath NHS Trust (Other); Gloucestershire Hospitals NHS Foundation Trust (Other); University Hospitals Bristol and Weston NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 3344; 2014-001948-37 (EudraCT Number)
Record Dates: First submitted 2014-07-25; First posted 2014-08-15 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-08

CONDITIONS: Post Partum Haemorrhage
Keywords: Post partum haemorrhage; Active Management of Third Stage of Labour; Carbetocin; Syntocinon; Syntometrine; Birth experience; Labour
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — carbetocin; Oxytocin; syntometrine; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Carbetocin (Experimental): One dose of 100 micrograms intramuscular Carbetocin given for active management of the third stage of labour, immediately after the birth of the baby
  Interventions: Drug: Carbetocin
- Syntocinon (Active Comparator): One dose of 10 International Units intramuscular Syntocinon given for active management of the third stage of labour, immediately after the birth of the baby
  Interventions: Drug: Syntocinon
- Syntometrine (Active Comparator): One dose of 500micrograms/5 International Units intramuscular Syntometrine given for active management of the third stage of labour, immediately after the birth of the baby
  Interventions: Drug: Syntometrine

INTERVENTIONS:
Drug: Carbetocin — The intervention is the administration of one dose of study drug to the recruited patient at the time of delivery. Carbetocin, listed here, is one of the of the three study drugs.
  Other Names: Pabal
  Arms: Carbetocin
Drug: Syntocinon — The intervention is the administration of one dose of study drug to the recruited patient at the time of delivery. Syntocinon, listed here, is one of the of the three study drugs.
  Other Names: Oxytocin
  Arms: Syntocinon
Drug: Syntometrine — The intervention is the administration of one dose of study drug to the recruited patient at the time of delivery. Syntometrine, listed here, is one of the of the three study drugs.
  Other Names: Syntometrine 500 micrograms/5 IU Solution for Injection
  Arms: Syntometrine

SUMMARY:
A quarter of all pregnancy and child-birth related deaths are due to excessive bleeding after the birth, "post-partum haemorrhage" (PPH). In the UK, PPH affects approx 10% of new mothers. PPH can be frightening for women and cause them to need additional treatments prolonging their hospital stay.

Commonly PPH is caused by an inadequately contracted womb after childbirth. Giving the mother an injection of "uterotonic" medicine following the birth of their baby can prevent this. It reduces the risk of PPH by 66%.

In the UK, the two medicines most commonly used are Syntocinon and Syntometrine. Syntometrine is longer acting, but a published review of trials concluded that Syntometrine is no better at preventing severe blood loss. Syntometrine is associated with more side effects including nausea, vomiting, and high blood pressure, and has been linked with rare, but fatal, cases of stroke. All guidelines therefore recommend Syntocinon for preventing PPH.Following a telephone survey of all maternity units in the UK, 71.4% of units still routinely use Syntometrine.

Carbetocin is a newer medicine, already widely used after caesarean section, but not yet after vaginal birth. Other studies have shown that Carbetocin is slightly better at preventing bleeding after birth when compared to Syntometrine, has fewer side effects than Syntometrine, and that it may be just as good as Syntocinon at preventing PPH. No studies have directly compared all three medicines or compared their overall cost; information vital to the NHS.

Investigators propose a trial of 5712 women over 13 months, in four maternity units to compare the effectiveness, side effects and cost of Syntocinon, Syntometrine and Carbetocin, for women having a vaginal birth.

Women will be randomly allocated to receive one of these drugs. Women and staff will not know which drug they receive. Staff will collect data such as the number of extra drugs and treatments needed and the volume of blood lost. Women will be asked to complete a side effects questionnaire. Investigators will perform an analysis of cost effectiveness once all results are available.

Aim: To directly compare the effectiveness, side effects and cost of Syntocinon, Syntometrine and Carbetocin given intramuscularly to prevent PPH in the 3rd stage of labour.

DETAILED DESCRIPTION:
BACKGROUND Around a quarter of all global pregnancy and child-birth related deaths are due to excessive bleeding after the birth of the baby and placenta, or "post-partum haemorrhage" (PPH). In the UK, PPH affects approximately 10% of new mothers. PPH can be extremely frightening for women and can cause them to need additional treatments including blood transfusion and removal of the womb as well as prolonging their hospital stay.

The most common cause of PPH is an inadequately contracted womb after childbirth. Giving the mother an injection of "uterotonic" medicine following the birth of their baby can prevent this. It reduces the risk of PPH by 66% and this should routinely be offered to all labouring women.

In the UK, the two medicines most commonly used for this purpose are Syntocinon and Syntometrine. Both mimic natural hormones. Syntometrine is longer acting, but a published review of trials comparing these two medicines concluded that Syntometrine is no better at preventing severe blood loss. Syntometrine is associated with more side effects including nausea, vomiting, and high blood pressure, and has been linked with rare, but fatal, cases of stroke. All guidelines therefore recommend Syntocinon for preventing PPH.

Our group conducted a telephone survey of all maternity units in the UK, and found that 71.4% of units still routinely use Syntometrine. Investigators estimate that 40,000-70,000 women per year are experiencing distressing nausea and vomiting in the emotionally important first few hours following childbirth. These women are also receiving a medicine with the potential to cause dangerous high blood pressure.

Carbetocin is a newer medicine, already widely used after caesarean section, but not yet after vaginal birth. Other studies have shown that Carbetocin is slightly better at preventing bleeding after birth when compared to Syntometrine, that it has fewer side effects than Syntometrine, and that it may be just as good as Syntocinon at preventing PPH. No studies have directly compared all three medicines or compared their overall cost; information vital to the NHS.

METHOD Investigators propose a trial of 5712 women over 13 months, in four maternity units in the South-West to compare the effectiveness, side effects and cost of Syntocinon, Syntometrine and Carbetocin, for women having a vaginal birth.

Women will be randomly allocated to receive one of these drugs. Women and staff will not know which drug they receive, so as not to influence the results collected. Staff will collect data such as the number of extra drugs and treatments needed and the volume of blood lost. Women will be asked to complete a side effects questionnaire. Investigators will perform an analysis of cost effectiveness once all results are available.

AIMS To directly compare the effectiveness, side effects and cost of Syntocinon, Syntometrine and Carbetocin given intramuscularly to prevent PPH in the 3rd stage of labour.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age at time of delivery
* Singleton pregnancy
* Vaginal birth (spontaneous and instrumental)
* >24 weeks gestation

Exclusion Criteria:

* Significant APH (>50ml) or suspected or proven placenta abruption
* Maternal coagulation disorder
* Intrauterine fetal death
* Patients who would decline blood products if required
* Known or suspected hypertensive disorders, including pre-eclampsia, pregnancy induced hypertension, essential hypertension (even if blood pressure well controlled)
* Hypertension in labour, or patients who have not had their blood pressure checked in labour
* Patients with peripheral, hepatic or cardiac disease
* Patients with an allergy or hypersensitivity to any of the active ingredients in Carbetocin, Syntometrine or Syntocinon
* Epilepsy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5798 (Actual)
Dates: Start 2015-02; Primary Completion 2018-08-31 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Requirement for additional uterotonic drugs within 24 hours of birth | From administration of prophylactic uterotonic agent to discharge from labour ward, within an expected average of 6 hours.
  Proportion of patients requiring additional uterotonic drugs after administration of study drug

SECONDARY OUTCOMES:
Estimated volume of blood loss at delivery | Within 24 hours of delivery
  Estimated volume of blood loss at delivery
Transfusion of blood products (type and number of units given) | From delivery until transfer from Labour Ward, within an expected average of 6 hours.
  Number of units of blood transfused, or volume of own blood returned to patient if intraoperative cell salvage used
Manual removal of placenta in theatre | From delivery until transfer from Labour Ward
  The requirement for the placenta to be removed in theatre
Requirement for surgical intervention to manage PPH | From delivery until transfer from Labour Ward, within an expected average of 2 days
  As a result of significant PPH a surgical intervention was required to manage the PPH
Maternal hypertension | First two postnatal hours following administration of study drug
  Hypertension
Maternal hypotension | In first two postnatal hours
  BP <90/60
Maternally-reported health-related quality of life | 24 hours after delivery and 14 days after delivery
  health-related quality of life reported by mother
Abdominal pain in the first two postnatal hours, recorded in Case Report Form (CRF) by midwife | First 2 post natal hours
  Patient reported secondary outcome
Post-partum vomiting | First 2 post natal hours
  Patient reported secondary outcome
Need for anti-emetic | First 2 post natal hours
  Patient reported secondary outcome
  By definition, labour starts when the patient is at least 3-4cm dilated with regular, painful contractions.
Headache | First two post natal hours
  Patient reported secondary outcome
Maternal experience of side effects | In first two post natal hours
  Captured using maternal side effects questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Tim Draycott, BMBS, Study Director — North Bristol NHS Trust/University of Bristol; Helen van der Nelson, BMBS, Study Chair — North Bristol NHS Trust/University of Bristol
Locations (5):
- United Kingdom (5):
  - North Bristol NHS Trust, Bristol, Avon
  - Gloucestershire Hospitals NHS Trust, Gloucester, Gloucestershire
  - Royal United Hospital NHS Trust, Bath, Somerset
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Great Western Hospital, Swindon

REFERENCES:
- [Derived] van der Nelson H, O'Brien S, Lenguerrand E, Marques E, Alvarez M, Mayer M, Burnard S, Siassakos D, Draycott T. Intramuscular oxytocin versus oxytocin/ergometrine versus carbetocin for prevention of primary postpartum haemorrhage after vaginal birth: study protocol for a randomised controlled trial (the IMox study). Trials. 2019 Jan 3;20(1):4. doi: 10.1186/s13063-018-3109-2. PMID 30606246